CLINICAL TRIAL: NCT01391494
Title: A Phase I Clinical Trial for Inactivated Enterovirus Type 71 Vaccine (Human Diploid Cell, KMB-17 Cell) in Chinese Adults, Children and Infants
Brief Title: A Safety Study of Inactivated EV71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Adults, Children and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EV71-KMB17-I-IMB-CAMS
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Human Enterovirus 71 (EV71); Hand, Foot and Mouth Disease; Inactivated Vaccine; Human Diploid cell; Safety; Immunogenicity; Adverse reactions associated with vaccine
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- 160Eu/0.5ml in adults (Experimental): inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 12 adults aged 18-49 years old on day 0, 14.
  Interventions: Biological: 160Eu/0.5ml in adults
- 320Eu/0.5ml in adults (Experimental): inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 12 adults aged 18-49 years old on day 0, 14.
  Interventions: Biological: 320Eu/0.5ml in adults
- 640Eu/0.5ml in adults (Experimental): inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 12 adults aged 18-49 years old on day 0, 14.
  Interventions: Biological: 640Eu/0.5ml in adults
- 1280Eu/0.5ml (without adjuvant) in adults (Experimental): inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 12 adults aged 18-49 years old on day 0, 14.
  Interventions: Biological: 1280Eu/0.5ml (without adjuvant) in 12 adults
- 0Eu/0.5ml in adults (Placebo Comparator): 0Eu/0.5ml placebo in 24 adults aged 18-49 years old on day 0, 14.
  Interventions: Biological: 0Eu/0.5ml in adults
- 160Eu/0.5ml in children (Experimental): inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 12 children aged 3-11 years old on day 0, 14.
  Interventions: Biological: 160Eu/0.5ml in children
- 320Eu/0.5ml in children (Experimental): inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 12 children aged 3-11 years old on day 0, 14.
  Interventions: Biological: 320Eu/0.5ml in children
- 640Eu/0.5ml in children (Experimental): inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 12 children aged 3-11 years old on day 0, 14.
  Interventions: Biological: 640Eu/0.5ml in children
- 1280Eu/0.5ml (without adjuvant) in children (Experimental): inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 12 children aged 3-11 years old on day 0, 14.
  Interventions: Biological: 1280Eu/0.5ml (without adjuvant) in children
- 0Eu/0.5ml in children (Placebo Comparator): 0Eu/0.5ml placebo in 24 children aged 3-11 years old on day 0, 14.
  Interventions: Biological: 0Eu/0.5ml in children
- 160Eu/0.5ml in infants (Experimental): inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 24 infants aged 6-35 months old on day 0, 28.
  Interventions: Biological: 160Eu/0.5ml in infants
- 320Eu/0.5ml in infants (Experimental): inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 24 infants aged 6-35 months old on day 0, 28.
  Interventions: Biological: 320Eu/0.5ml in infants
- 640Eu/0.5ml in infants (Experimental): inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 24 infants aged 6-35 months old on day 0, 28.
  Interventions: Biological: 640Eu/0.5ml in infants
- 1280Eu/0.5ml (without adjuvant) in infants (Experimental): inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 24 infants aged 6-35 months old on day 0, 28.
  Interventions: Biological: 1280Eu/0.5ml (without adjuvant) in infants
- 0Eu/0.5ml in infants (Placebo Comparator): 0Eu/0.5ml placebo in 48 infants aged 6-35 months old on day 0, 28.
  Interventions: Biological: 0Eu/0.5ml in infants

INTERVENTIONS:
Biological: 160Eu/0.5ml in adults — inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 12 adults aged 18-49 years old on day 0, 14.
  Arms: 160Eu/0.5ml in adults
Biological: 320Eu/0.5ml in adults — inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 12 adults aged 18-49 years old on day 0, 14.
  Arms: 320Eu/0.5ml in adults
Biological: 640Eu/0.5ml in adults — inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 12 adults aged 18-49 years old on day 0, 14.
  Arms: 640Eu/0.5ml in adults
Biological: 1280Eu/0.5ml (without adjuvant) in 12 adults — inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 12 adults aged 18-49 years old on day 0, 14.
  Arms: 1280Eu/0.5ml (without adjuvant) in adults
Biological: 0Eu/0.5ml in adults — 0Eu/0.5ml placebo in 24 adults aged 18-49 years old on day 0, 14.
  Arms: 0Eu/0.5ml in adults
Biological: 160Eu/0.5ml in children — inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 12 children aged 3-11 years old on day 0, 14.
  Arms: 160Eu/0.5ml in children
Biological: 320Eu/0.5ml in children — inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 12 children aged 3-11 years old on day 0, 14.
  Arms: 320Eu/0.5ml in children
Biological: 640Eu/0.5ml in children — inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 12 children aged 3-11 years old on day 0, 14.
  Arms: 640Eu/0.5ml in children
Biological: 1280Eu/0.5ml (without adjuvant) in children — inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 12 children aged 3-11 years old on day 0, 14.
  Arms: 1280Eu/0.5ml (without adjuvant) in children
Biological: 0Eu/0.5ml in children — 0Eu/0.5ml placebo in 24 children aged 3-11 years old on day 0, 14.
  Arms: 0Eu/0.5ml in children
Biological: 160Eu/0.5ml in infants — inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 24 infants aged 6-35 months old on day 0, 28.
  Arms: 160Eu/0.5ml in infants
Biological: 320Eu/0.5ml in infants — inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 24 infants aged 6-35 months old on day 0, 28.
  Arms: 320Eu/0.5ml in infants
Biological: 640Eu/0.5ml in infants — inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 24 infants aged 6-35 months old on day 0, 28.
  Arms: 640Eu/0.5ml in infants
Biological: 1280Eu/0.5ml (without adjuvant) in infants — inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 24 infants aged 6-35 months old on day 0, 28.
  Arms: 1280Eu/0.5ml (without adjuvant) in infants
Biological: 0Eu/0.5ml in infants — 0Eu/0.5ml placebo in 48 infants aged 6-35 months old on day 0, 28.
  Arms: 0Eu/0.5ml in infants

SUMMARY:
Enterovirus 71 (EV71), a major pathogen that is responsible for causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae.

Since the late 1990s, a series of large HFMD epidemics caused by EV71 have been reported in the Asia-Pacific region. Notably, there is evidence that the most severe cases from these epidemic outbreaks are associated with neurological disorders with CNS involvement caused by EV71 infection. Because of these EV71 infection-related public health issues, the research and development of EV71 vaccine candidates have been heavily promoted.

Recently, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, including inactivated vaccine, attenuated vaccine, subunit vaccine, DNA vaccine, epitope peptide vaccine, virus-like particles (VLPs).

Basing on the previous studies of elicited protection in mice and rhesus monkeys, a formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been licensed by SFDA in China, Dec. 2010. The phase I clinical trial has been carried out, during four months, in Guangxi Province, China. The purpose of this study is to evaluate the safety, tolerability and immunogenicity of the formalin-inactivated EV71 vaccine in Chinese adults (from 18 to 49 years old), children (from 3 to 11 years old) and infants (from 6 to 35 months old).

DETAILED DESCRIPTION:
Hand-foot-and-mouth disease (HFMD) is a significant cause of death, usually characterized by vesicular lesions on the skin and oral mucosa and high morbidity rates in children. Additionally, occasional fatal cases have been reported involving brainstem encephalitis and myelitis associated with cardiopulmonary collapse. Pulmonary edema/hemorrhage and respiratory failure are the major causes of death among children less than five years old.

Enterovirus 71 (EV71), a major pathogen that is responsible for causing HFMD worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Since the late 1990s, a series of large HFMD epidemics caused by EV71 have been reported in the Asia-Pacific region. Notably, there is evidence that the most severe cases from these epidemic outbreaks are associated with neurological disorders with CNS involvement caused by EV71 infection. Because of these EV71 infection-related public health issues, the research and development of EV71 vaccine candidates have been heavily promoted.

Recently, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, including heat-inactivated or formalin-inactivated vaccine, live-attenuated vaccine, recombinant viral protein 1 (VP1) vaccine, VP1 DNA vaccine, VP1 epitope peptide vaccine, EV71 virus-like particles (VLPs) and bacterial or viral vector expressing VP1. Overall, the inactivated whole-virus vaccines seem to be more immunogenic than recombinant VP1 and DNA vaccines.

Basing on the previous studies of elicited protection in mice and rhesus monkeys (Ying Zhang, et al. Pathogenesis study of Enterovirus 71 Infection in Rhesus Monkeys. Lab Invest, 2011, doi:10.1038/labinest.2011.82; Longding Liu, et al. Neonatal Rhesus Monkey is a Potential Animal Model for Studying Pathogenesis of EV71 Infection. Virology, 2011, 412:91-100; Chenghong Dong, et al. Immunoprotection Elicited by an Enterovirus Type 71 Experimental Inactivated Vaccine in Mice and Rhesus Monkeys. Vaccine, 2011, doi: 10.1016/j.vaccine.2011.06.044.), a formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been licensed by SFDA in China, Dec. 2010. The phase I clinical trial has been carried out, during four months, in Guangxi Province, China. The purpose of this study is to evaluate the safety, tolerability and immunogenicity of the formalin-inactivated EV71 vaccine in Chinese adults (from 18 to 49 years old), children (from 3 to 11 years old) and infants (from 6 to 35 months old).

ELIGIBILITY:
For the subjects aged from 18-49 years old adults:

Inclusion Criteria:

* Healthy subjects (18-49 years old adults) as established by medical history and clinical examination
* The subjects oneself or their legal guardian must be aware of this vaccines
* Voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0℃
* With the ability and objective to comply with the requirements of the protocol
* Persist for a 2-month visit and receive blood tests according to program requirements

Exclusion Criteria:

* Subject who has a clinical diagnosis history of Hand, Foot and Mouth Disease (HFMD)
* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Severe malnutrition or dysgenopathy
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 28 days or 1 months
* Any prior administration of subunit or inactivated vaccines in last 14 days
* Under the anti-TB prevention or therapy
* Fever before vaccination, axillary temperature ﹥37.0℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140mmHg and/or diastolic blood pressure ﹥90mmHg; systolic blood pressure ﹤90mmHg and/or diastolic blood pressure ﹤60mmHg
* Breast-feeding, pregnant, planning a pregnancy within 60 days or positive pregnancy test women
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

For the subjects aged from 3-11 years old children:

Inclusion Criteria:

* Healthy subjects (3-11 years old children) as established by medical history and clinical examination
* Full-term (37-42 weeks), weight ≥ 2500 g when it was born
* The subjects' legal guardian must be aware of this vaccines
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0℃
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol
* Persist for a 2-month visit and receive blood tests according to program requirements

Exclusion Criteria:

* Subject who has a clinical diagnosis history of Hand, Foot and Mouth Disease (HFMD)
* ≤37 weeks gestation
* weight ≤ 2500 g when it was born
* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Severe malnutrition or dysgenopathy
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 28 days or 1 months
* Any prior administration of subunit or inactivated vaccines in last 14 days
* Under the anti-TB prevention or therapy
* Fever before vaccination, axillary temperature ﹥37.0℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140mmHg and/or diastolic blood pressure ﹥90mmHg; systolic blood pressure ﹤90mmHg and/or diastolic blood pressure ﹤60mmHg
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

For the subjects aged from 6-35 months infants:

Inclusion Criteria:

* Healthy subjects (6-35 months infants) as established by medical history and clinical examination
* Full-term (37-42 weeks), weight ≥ 2500 g when it was born
* The subjects' legal guardian must be aware of this vaccines
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0℃
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol
* Persist for a 2-month visit and receive blood tests according to program requirements

Exclusion Criteria:

* Subject who has a clinical diagnosis history of Hand, Foot and Mouth Disease (HFMD)
* ≤37 weeks gestation
* weight ≤ 2500 g when it was born
* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Severe malnutrition or dysgenopathy
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 28 days or 1 months
* Any prior administration of subunit or inactivated vaccines in last 14 days
* Under the anti-TB prevention or therapy
* Fever before vaccination, axillary temperature ﹥37.0℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140mmHg and/or diastolic blood pressure ﹥90mmHg; systolic blood pressure ﹤90mmHg and/or diastolic blood pressure ﹤60mmHg
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 288 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the Safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Adults. | within the first 14 days after the first vaccination
  Adverse reactions associated with vaccine were observed in Chinese Adults (from 18 to 49 years old) after the first vaccination.
Evaluate the Safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Adults. | within the first 4 days after the second vaccination
  Adverse reactions associated with vaccine were observed in Chinese Adults (from 18 to 49 years old) after the second vaccination.
Evaluate the Safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Children. | within the first 14 days after the first vaccination
  Adverse reactions associated with vaccine were observed in Chinese Children (from 3 to 11 years old) after the first vaccination.
Evaluate the Safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Children. | within the first 4 days after the second vaccination
  Adverse reactions associated with vaccine were observed in Chinese Children (from 3 to 11 years old) after the second vaccination.
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants. | within the first 28 days after the first vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants (from 6 to 35 months old) after the first vaccination.
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants. | within the first 28 days after the second vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants (from 6 to 35 months old) after the second vaccination.

SECONDARY OUTCOMES:
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of adults, children and infant, after first vaccination. | within the first 14 or 28 days after the first vaccination
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of adults within the first 14 days after first vaccination.
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of children within the first 14 days after first vaccination.
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of infant, within the first 28 days after first vaccination.
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of adults, children and infant, after second vaccination. | within the first 4 or 28 days after the second vaccination
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of adults within the first 4 days after second vaccination.
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of children within the first 4 days after second vaccination.
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of infant, within the first 28 days after second vaccination.
Evaluate the seroconversion rate of antinuclear antibodies in serum of adults, children and infant, after first vaccination. | within the first 14 or 28 days after the first vaccination
  The seroconversion rate of antinuclear antibodies was evaluated in serum of adults within the first 14 days after first vaccination.
  The seroconversion rate of antinuclear antibodies was evaluated in serum of children within the first 14 days after first vaccination.
  The seroconversion rate of antinuclear antibodies was evaluated in serum of infant, within the first 28 days after first vaccination.
Evaluate the seroconversion rate of antinuclear antibodies in serum of adults, children and infant, after second vaccination. | within the first 4 or 28 days after the second vaccination
  The seroconversion rate of antinuclear antibodies was evaluated in serum of adults within the first 4 days after the second vaccination.
  The seroconversion rate of antinuclear antibodies was evaluated in serum of children within the first 4 days after the second vaccination.
  The seroconversion rate of antinuclear antibodies was evaluated in serum of infant, within the first 28 days after the second vaccination.
Evaluate the abnormity change of live and kidney function indexes in serum of adults, children and infant, after first vaccination. | within the first 14 or 28 days after the first vaccination
  The abnormity change of live and kidney function indexes were evaluated in serum of adults within the first 14 days after first vaccination.
  The abnormity change of live and kidney function indexes were evaluated in serum of children within the first 14 days after first vaccination.
  The abnormity change of live and kidney function indexes were evaluated in serum of infant, within the first 28 days after first vaccination.
Evaluate the abnormity change of live and kidney function indexes in serum of adults, children and infant, after second vaccination. | within the first 4 or 28 days after the second vaccination
  The abnormity change of live and kidney function indexes were evaluated in serum of adults within the first 4 days after the second vaccination.
  The abnormity change of live and kidney function indexes were evaluated in serum of children within the first 4 days after the second vaccination.
  The abnormity change of live and kidney function indexes were evaluated in serum of infant, within the first 28 days after the second vaccination.
Evaluate the vaccine-induced cellular immune responses in infant after first vaccination. | within the first 28 days after the first vaccination
  The vaccine-induced cellular immune responses were evaluated in serum of infant, within the first 28 days after the first vaccination.
Evaluate the vaccine-induced cellular immune responses in infant after second vaccination. | within the first 28 days after the second vaccination
  The vaccine-induced cellular immune responses were evaluated in serum of infant, within the first 28 days after the second vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Master, Principal Investigator — Guangxi Provincial Center for Diseases Control and Prevention
Locations (1):
- Guangxi Provincial Center for Diseases Control and Prevention, Nanning, Guangxi, China

REFERENCES:
- [Derived] Liu L, Zhang Y, Wang J, Zhao H, Jiang L, Che Y, Shi H, Li R, Mo Z, Huang T, Liang Z, Mao Q, Wang L, Dong C, Liao Y, Guo L, Yang E, Pu J, Yue L, Zhou Z, Li Q. Study of the integrated immune response induced by an inactivated EV71 vaccine. PLoS One. 2013;8(1):e54451. doi: 10.1371/journal.pone.0054451. Epub 2013 Jan 23. PMID 23372725
- See also: The rhesus monkey model may be used to study not only the basic pathogenesis of EV71 viral infections, but also to examine clinical features, such as neurological lesions, in the CNS and pathological changes in associated organs. — http://www.nature.com/labinvest/journal/vaop/ncurrent/abs/labinvest201182a.html